CLINICAL TRIAL: NCT06633081
Title: Smartphone Addiction and Isometric Rotator Cuff Muscles Strength Among Adults
Brief Title: Smartphone Addiction and Isometric Strength of Rotator Cuff Muscles
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Abdallah Mohamed Bashier, Principal Investigator, Cairo University
Other Study IDs: REC/PT/012/0167
Record Dates: First submitted 2024-09-27; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: handheld dynamometer — handheld dynamometer is a device that measure muscle strength

SUMMARY:
To investigate the relationship between smartphone addiction and isometric rotator cuff muscles strength among adults

DETAILED DESCRIPTION:
Smartphones play an important role in human life because they are used for communication, accessing the internet, and gaming. The rate of smartphone usage has increased over the last decade, as has the duration and frequency of use. according to one study, 79 percent of people aged 18 to 44 spent almost all of their time on their smartphones, with only two hours of the day spent without one.

No previous study has found a link between smartphone addiction and isometric Rotator Cuff muscular strength, to the authors' knowledge. Therefore, the primary purpose of this study will be to determine the relationship between smartphone addiction and isometric rotator cuff muscles strength.

ELIGIBILITY:
Inclusion Criteria:

- 1- This study will comprise healthy volunteers between the ages of 18 and 30 who needed to use a smart phone.

2- Subjects who put in more than 4 hours per day using smartphone.

Exclusion Criteria:

* Patients will rule out if

  1. They had any medical condition that could cause shoulder pain (such as impingement, subacromial bursitis, rotator cuff damage, or traumatic or degenerative supraspinatus tendonitis).
  2. Anyone with a positive Neer sign, a positive Hawkins sign, discomfort during shoulder elevation, pain at the location of the rotator cuff tendon, pain with resisted isometric shoulder abduction, or a history of pain in the C5 dermatome will be ruled out.
  3. Any individual who had previously suffered a musculoskeletal injury or surgery that could have influenced the measurement will be also eliminated.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1- This study will comprise 300 healthy volunteers between the ages of 18 and 30 who needed to use a smart phone
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
isometric strength of rotator cuff | up to 3 month
  Hand-held Dynamometer (HHD) is an ergonomic hand-held device used for objectively quantifying muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic, faculty of Physical Therapy Cairo University, Giza, Giza Governorate, Egypt

REFERENCES:
- [Background] Ergun Kesli E, Guclu B, Ozden F, Dilek B. Investigation of grip strength, pain threshold, pain tolerance and function in smartphone users. Somatosens Mot Res. 2023 Sep;40(3):103-109. doi: 10.1080/08990220.2023.2186392. Epub 2023 Mar 13. PMID 36908251
- [Background] Alshahrani A, Samy Abdrabo M, Aly SM, Alshahrani MS, Alqhtani RS, Asiri F, Ahmad I. Effect of Smartphone Usage on Neck Muscle Endurance, Hand Grip and Pinch Strength among Healthy College Students: A Cross-Sectional Study. Int J Environ Res Public Health. 2021 Jun 10;18(12):6290. doi: 10.3390/ijerph18126290. PMID 34200762
- [Background] Ratan ZA, Parrish AM, Zaman SB, Alotaibi MS, Hosseinzadeh H. Smartphone Addiction and Associated Health Outcomes in Adult Populations: A Systematic Review. Int J Environ Res Public Health. 2021 Nov 22;18(22):12257. doi: 10.3390/ijerph182212257. PMID 34832011